CLINICAL TRIAL: NCT06051084
Title: Advancing Our Understanding and Treatment of Anxiety Through Bringing Together Facets of Conscious Experience and Brain Mechanisms: Open/Closed Meets the Default Mode Network
Brief Title: Investigating How the Brain Processes Different Experiences
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Dartmouth College (Other); Tiny Blue Dot Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022003264
Record Dates: First submitted 2023-09-18; First posted 2023-09-22 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Anxiety
Keywords: Anxiety; Mindfulness; MRI; Cell Phone
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App-Delivered Mindfulness Training (MT) (Experimental): The program is delivered via a smartphone-based platform, which includes a progression through 30+ daily modules of brief didactic and experience-based mindfulness training (videos and animations), app-triggered check-ins to encourage engagement, and user-initiated guided mindfulness exercises to help disrupt worry cycles in the moment.
  Interventions: Behavioral: App-Delivered Mindfulness Training (MT)
- App-Delivered Coloring (Active Comparator): An app-based coloring book with a variety of designs to choose from including mandalas, animal patterns, and florals. It is designed to help individuals relax and reduce stress and anxiety based on the benefits found in past research studies.
  Interventions: Behavioral: App-Delivered Coloring

INTERVENTIONS:
Behavioral: App-Delivered Mindfulness Training (MT) — The program is delivered via a smartphone-based platform, which includes a progression through 30+ daily modules of brief didactic and experience-based mindfulness training (videos and animations), app-triggered check-ins to encourage engagement, and user-initiated guided mindfulness exercises to help disrupt worry cycles in the moment.
  Arms: App-Delivered Mindfulness Training (MT)
Behavioral: App-Delivered Coloring — An app-based coloring book with a variety of designs to choose from including mandalas, animal patterns, and florals. It is designed to help individuals relax and reduce stress and anxiety based on the benefits found in past research studies.
  Arms: App-Delivered Coloring

SUMMARY:
The goal of this clinical trial is to test the efficacy of an app-based program in reducing anxiety and exploring associated changes in brain activity.

DETAILED DESCRIPTION:
The main question[s] it aims to answer are:

PRIMARY AIM: Confirm that the conscious experience of open/closed correlates with P/PCC activation/deactivation.

SECONDARY AIM: Determine if changes in P/PCC activity predict clinical outcomes (GAD-7 scores) in individuals with moderate to severe anxiety after using an app.

Participants may be asked to:

* Complete a Zoom interview
* Complete online surveys at baseline and 2 months post-treatment initiation
* Complete MRIs at baseline and 2 months post-treatment initiation
* Wear a smartwatch and answer daily questions about their anxiety
* Use an app daily

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 65 years
2. Able to travel to Brown University for research assessment
3. Able to speak English because all study activities will be conducted in English.
4. GAD-7 ≥ 10
5. Owns a smartphone

Exclusion Criteria:

1. If using psychotropic medication - not on a stable dosage at least 6 weeks
2. As needed (i.e., prn) benzodiazepine use
3. Psychotic disorder (e.g., bipolar disorder, schizophrenia, schizoaffective disorder, psychosis)
4. MRI contraindications
5. Claustrophobia
6. Recreational drug use past 2 weeks
7. Alcohol abuse
8. Pregnancy or plans to become pregnant
9. Cohabiting with a study participant
10. Weight ≥ 300 lbs (due to inability to fit in scanner)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in GAD - 7 | collected at baseline and 2 month follow up apt
  Generalized Anxiety Disorder 7-items (GAD-7). The GAD-7 is a validated 7-item measure of anxiety rated on a 4-point Likert scale ranging from 0 (Not at all sure) to 3 (Nearly every day).
Change From Baseline in Posterior Cingulate Cortex (PCC) Blood Oxygen Level Dependent (BOLD) Signal | collected at baseline and 2 month follow up apt
  BOLD signal change will be measured by fMRI and analyzed using statistical parametric mapping

SECONDARY OUTCOMES:
Penn State Worry Questionnaire (PSWQ) | collected at baseline and 2 month follow up apt
  The PSWQ is a validated 16-item self-report measure of worry with items presented on a 5-point Likert scale ranging from 1 (not at all typical of me) to 5 (very typical of me).
Five Facet Mindfulness Questionnaire (FFMQ) non-reactivity scale | collected at baseline and 2 month follow up apt
  The non-reactivity scale is a validated subscale of the 39-item FFMQ which is a self-report psychological measure of mindfulness skills. This subscale contains 7 items which are presented on a 6-point Likert scale ranging from 1 (almost always) to 6 (almost never).

OTHER OUTCOMES:
Multidimensional Assessment of Interoceptive Awareness (MAIA) | collected at baseline and 2 month follow up apt
  The MAIA is a validated 32-item self-report questionnaire comprised of 8 subscales including: noticing, not-distracting, not-worrying, attention regulation, emotional awareness, self-regulation, body listening, and trusting. Items are rated on a 6-point Likert scale ranging from 0 (never) to 5 (always).
Anxiety Sensitivity Index (ASI) | collected at baseline and 2 month follow up apt
  The ASI is a validated 16-item self-report measure of the fear of anxiety sensations. Items are rated on a 5-point Likert scale ranging from 0 (Very little) to 4 (Very much).
Interest (I) Type and Deprivation (D) Type scale (I/D) | collected at baseline and 2 month follow up apt
  The I/D scale is a validated 10-item self-report measure of curiosity. Items are rated on a 4-point Likert scale ranging from 1 (Almost never) to 4 (Almost always).
Acceptance & Action questionnaire (AAQ-II) | collected at baseline and 2 month follow up apt
  The AAQ-II is a validated 7-item self-report measure of experiential avoidance. Items are rated on a 7-point Likert scale ranging from 1 (Never true) to 7 (Always true).
Intolerance of Uncertainty 12-item scale (IUS-12) | collected at baseline and 2 month follow up apt
  The IUS-12 is a validated 12-item self-report measure of intolerance of uncertainty. Items are rated on a 5-point Likert scale ranging from 1 (Not at all characteristic of me) to 5 (Entirely characteristic of me).

CONTACTS AND LOCATIONS:
Overall Officials: Judson Brewer, MD, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No